CLINICAL TRIAL: NCT01417000
Title: A Phase 2, Randomized, Multicenter, Open-Label Study of the Efficacy and Immune Response of the Sequential Administration of GVAX Pancreas Vaccine Alone or Followed by CRS-207 in Adults With Metastatic Pancreatic Adenocarcinoma
Brief Title: Safety and Efficacy of Combination Listeria/GVAX Immunotherapy in Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aduro Biotech, Inc. (Industry)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ADU-CL-01; NCT01468870 (obsolete NCT alias)
Record Dates: First submitted 2011-08-10; First posted 2011-08-16 (Estimated); Results first posted 2018-05-08 (Actual); Last update posted 2018-05-08 (Actual); Status verified 2018-04

CONDITIONS: Metastatic Pancreatic Cancer
Keywords: Cancer; Cancer vaccine; Listeria monocytogenes; Listeria-based vaccines; GVAX; Cyclophosphamide; Cytoxan; T regulatory cells; Heterologous Prime-Boost; Immunotherapy; Mesothelin; Pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasms | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cy/GVAX + CRS-207 (Experimental): 200 mg per square meter (mg/m^2) cyclophosphamide (Cy) administered by intravenous (IV) infusion on Day 1 of Weeks 1 and 4; GVAX pancreas vaccine (GVAX, 5 × 10e8 cells) administered by intradermal injection on Day 2 of Weeks 1 and 4; CRS-207 (1 × 10e9 colony forming units [CFU]) administered by IV infusion on Day 1 of Weeks 7, 10, 13, 16.
  Interventions: Biological: GVAX Pancreas; Biological: CRS-207; Drug: Cyclophosphamide
- Cy/GVAX (Experimental): 200 mg/m^2 Cy administered by IV infusion on Day 1 of Weeks 1, 4, 7, 10, 13, 16; GVAX (5 × 10e8 cells) administered by intradermal injection on Day 2 of Weeks 1, 4, 7, 10, 13, 16.
  Interventions: Biological: GVAX Pancreas; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: GVAX Pancreas
  Other Names: GVAX
Biological: CRS-207
  Arms: Cy/GVAX + CRS-207
Drug: Cyclophosphamide
  Other Names: Cytoxan; Cy

SUMMARY:
Test the safety, immune response and efficacy of GVAX pancreas vaccine (with cyclophosphamide) and CRS-207 compared to GVAX pancreas vaccine (with cyclophosphamide) alone in adults who have failed or refused prior treatment for metastatic pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Have histologically proven malignant adenocarcinoma of the pancreas; measurable disease is not required. (Subjects with mixed histology will be included if the predominant component is adenocarcinoma. Subjects must have metastatic disease.)
* Have received or refused at least one chemotherapy regimen
* At least 18 years of age
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Anticipated life expectancy of >12 weeks
* For women and men of childbearing potential, a medically acceptable method of highly effective contraception (oral hormonal contraceptive, condom plus spermicide, or hormone implants) must be used throughout the study period and for 28 days after their final vaccine administration. (A barrier method of contraception must be employed by all subjects [male and female], regardless of other methods.)
* Be willing and able to give written informed consent, and be able to comply with all study procedures
* Have adequate organ function as defined by specified laboratory values

Exclusion Criteria:

* Currently have or have history of certain study-specified heart, liver, kidney, lung, neurological, immune or other medical conditions
* Known history or evidence of brain metastases
* Have any evidence of hepatic cirrhosis or clinical or radiographic ascites
* Have clinically significant and/or malignant pleural effusion
* Known or suspected hypersensitivity to any component of GVAX Pancreas vaccine or CRS-207, or known allergy to both penicillin and sulfa
* Received an investigational product within 28 days of study treatment or planned to receive within 28 days after vaccine administration
* Used any systemic steroids within 28 days of study treatment
* Use more than 3 g/d of acetaminophen
* Prosthetic joint or other artificial implant or device that cannot be easily removed (there are some exceptions)
* Major surgery or significant traumatic injury (or unhealed surgical wounds) occurring within 28 days prior to receiving study drug, or planned surgery requiring general anesthesia
* Infection with HIV or hepatitis B or C at screening
* Any immunodeficiency disease or immunocompromised state or active autoimmune disease or history of autoimmune disease requiring systemic steroids or other immunosuppressive treatment
* Be pregnant or breastfeeding
* Unable to avoid close contact with another individual known to be at high risk of listeriosis (e.g., newborn infant, pregnant woman, HIV-positive individual) during the course of CRS-207 treatment until completion of antibiotic regimen
* Conditions, including alcohol or drug dependence, intercurrent illness, or lack of sufficient peripheral venous access, that would affect the patient's ability to comply with study visits and procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2011-09-21 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2017-02-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dung T Le, MD, Principal Investigator — Johns Hopkins University
Locations (10):
- United States (10):
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins Hospital, Baltimore, Maryland
  - National Cancer Institute, Bethesda, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - NYU Langone Medical Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center of Columbia University, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Providence Portland Medical Center, Portland, Oregon
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Virginia Mason Medical Center, Seattle, Washington

REFERENCES:
- [Background] Brockstedt DG, Giedlin MA, Leong ML, Bahjat KS, Gao Y, Luckett W, Liu W, Cook DN, Portnoy DA, Dubensky TW Jr. Listeria-based cancer vaccines that segregate immunogenicity from toxicity. Proc Natl Acad Sci U S A. 2004 Sep 21;101(38):13832-7. doi: 10.1073/pnas.0406035101. Epub 2004 Sep 13. PMID 15365184
- [Background] Laheru D, Lutz E, Burke J, Biedrzycki B, Solt S, Onners B, Tartakovsky I, Nemunaitis J, Le D, Sugar E, Hege K, Jaffee E. Allogeneic granulocyte macrophage colony-stimulating factor-secreting tumor immunotherapy alone or in sequence with cyclophosphamide for metastatic pancreatic cancer: a pilot study of safety, feasibility, and immune activation. Clin Cancer Res. 2008 Mar 1;14(5):1455-63. doi: 10.1158/1078-0432.CCR-07-0371. PMID 18316569
- [Background] Le DT, Dubenksy TW Jr, Brockstedt DG. Clinical development of Listeria monocytogenes-based immunotherapies. Semin Oncol. 2012 Jun;39(3):311-22. doi: 10.1053/j.seminoncol.2012.02.008. PMID 22595054
- [Background] Le DT, Wang-Gillam A, Picozzi V, Greten TF, Crocenzi T, Springett G, Morse M, Zeh H, Cohen D, Fine RL, Onners B, Uram JN, Laheru DA, Lutz ER, Solt S, Murphy AL, Skoble J, Lemmens E, Grous J, Dubensky T Jr, Brockstedt DG, Jaffee EM. Safety and survival with GVAX pancreas prime and Listeria Monocytogenes-expressing mesothelin (CRS-207) boost vaccines for metastatic pancreatic cancer. J Clin Oncol. 2015 Apr 20;33(12):1325-33. doi: 10.1200/JCO.2014.57.4244. Epub 2015 Jan 12. PMID 25584002
- See also: For more information, please click here to visit Aduro's website. — http://www.aduro.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled subjects with malignant metastatic adenocarcinoma of the pancreas who had received or refused at least one prior chemotherapy regimen. Study was conducted in the United States at 10 medical centers; however, 1 center did not enroll any subjects. The last subject completed the study in February 2017.
Pre-assignment Details: Participants screened over a 28-day period.
Period: Overall Study
Arm/Group | Cy/GVAX + CRS-207 | Cy/GVAX
Started (Participant flow values reflect original arm assignments and do not account for rollover subjects) | 61 (62 subjects randomized into Cy/GVAX + CRS-207 arm; 61 subjects received ≥ 1 protocol-specified drug.) | 29 (31 subjects randomized into Cy/GVAX arm; 29 subjects received ≥ 1 protocol-specified drug.)
Completed (No predetermined study completion date or study completion event specified in protocol.) | 0 (Subjects followed until lost to follow-up/death/study close, so no subjects "completed" study.) | 0 (Subjects followed until lost to follow-up/death/study close, so no subjects "completed" study.)
Not Completed | 61 | 29
Not completed — Death | 59 | 28
Not completed — Lost to Follow-up | 1 | 0
Not completed — Study Terminated by Sponsor | 1 | 1

BASELINE CHARACTERISTICS:
Population: Baseline analysis provided for the Full Analysis Set (FAS), defined as those randomized study subjects who were administered at least 1 dose of protocol-specified drug. Baseline analysis is provided for subjects on the basis of their original study arm assignments, prior to any rollover from the Cy/GVAX arm to the Cy/GVAX + CRS-207 arm.
Groups:
- Cy/GVAX + CRS-207: 200 mg/m^2 Cy administered by IV infusion on Day 1 of Weeks 1 and 4; GVAX pancreas vaccine (5 × 10e8 cells) administered by intradermal injection on Day 2 of Weeks 1 and 4; CRS-207 (1 × 10e9 CFU) administered by IV infusion on Day 1 of Weeks 7, 10, 13, 16.
- Cy/GVAX: 200 mg/m^2 Cy administered by IV infusion on Day 1 of Weeks 1, 4, 7, 10, 13, 16; GVAX pancreas vaccine (5 × 10e8 cells) administered by intradermal injection on Day 2 of Weeks 1, 4, 7, 10, 13, 16.
- Total: Total of all reporting groups
Arm/Group | Cy/GVAX + CRS-207 | Cy/GVAX | Total
Number analyzed (Participants) | 61 | 29 | 90
Age, Continuous [Median (Standard Deviation); unit: years] | 63.7 (9.14) | 63.9 (9.29) | 63.8 (9.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 10 | 37
  Male | 34 | 19 | 53

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) in Subjects Receiving Test Treatments (FAS)
Description: For all treated subjects, OS was defined as the time between the date of randomization and the date of death or censoring, and was estimated using Kaplan-Meier (KM) methods with 95% confidence intervals (CIs). Subjects without documentation of death at the time of the final analysis were censored using the date the subject was last known to be alive. Per the study protocol, following an Interim Analysis (IA), subjects in the Cy/GVAX arm were offered rollover to Cy/GVAX + CRS-207 arm. 3 subjects rolled over to the Cy/GVAX + CRS-207 arm (rollover subjects). These rollover subjects were censored at the day prior to the first rollover treatment dose date, and were included for analysis in the Cy/GVAX arm. Additionally, 2 subjects originally treated per the Cy/GVAX + CRS-207 arm discontinued treatment and entered follow-up, but following IA were re-treated per the Cy/GVAX + CRS-207 arm regimen. Data from these "re-treated subjects" were included in the Cy/GVAX + CRS-207 arm analysis.
Time Frame: Subjects were followed from the date of randomization to the date of death or discontinuation, whichever came first, assessed up to 60 months.
Population: Analysis conducted for the FAS of each study arm.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cy/GVAX + CRS-207 | Cy/GVAX
Number analyzed (Participants) | 61 | 29
months | 6.28 [4.47 to 9.40] | 4.07 [3.32 to 5.42]

2. Secondary Outcome: To Assess Safety of the Cyclophosphamide, GVAX Pancreas Vaccine, and CRS-207 Treatment Regimen
Description: Safety was assessed based upon the number of adverse events (AEs) that occurred in the FAS of each treatment arm, including serious AEs and total AEs. Total AEs included both serious and non-serious AEs. AEs reported for the Cy/GVAX + CRS-207 arm (FAS) include the 61 treated subjects initially assigned to this arm plus AEs occurring on/after the first rollover dose date for the 3 Cy/GVAX rollover subjects. AEs reported for the Cy/GVAX arm (FAS) include treated subjects initially assigned to this arm but exclude AEs for rollover subjects occurring on/after the first rollover dose date.
Time Frame: Starting with administration of first investigational drug product through 28 days after final study treatment, assessed up to 60 months from the date of randomization.
Population: Analysis conducted for the FAS of each study arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Cy/GVAX + CRS-207 | Cy/GVAX
Number analyzed (Participants) | 64 | 29
Participants
  Serious AEs | 29 | 10
  Total AEs | 64 | 29

ADVERSE EVENTS:
Time Frame: Starting with administration of first investigational drug product through 28 days after final study treatment, assessed up to 60 months from the date of randomization.
Description: AEs reported for the Cy/GVAX + CRS-207 arm (FAS) include the 61 treated subjects initially assigned to this arm plus AEs occurring on/after the first rollover dose date for the 3 Cy/GVAX rollover subjects. AEs reported for the Cy/GVAX arm (FAS) include treated subjects initially assigned to this arm but exclude AEs for rollover subjects occurring on/after the first rollover dose date. AEs reported in the "Other (Not Including Serious) Adverse Events" section include serious and non-serious AEs.
Arm/Group | Cy/GVAX + CRS-207 | Cy/GVAX
Serious Adverse Events (participants affected / at risk) | 29/64 | 10/29
Other Adverse Events (participants affected / at risk) | 64/64 | 29/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cy/GVAX + CRS-207 (N=64) | Cy/GVAX (N=29)
OBSTRUCTION GASTRIC (Gastrointestinal disorders) | 4 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 3 | 0
ASCITES (Gastrointestinal disorders) | 2 | 0
DUODENAL OBSTRUCTION (Gastrointestinal disorders) | 1 | 0
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 | 0
INTESTINAL PERFORATION (Gastrointestinal disorders) | 1 | 0
NAUSEA (Gastrointestinal disorders) | 1 | 0
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 3 | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 3 | 1
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
CHOLANGITIS (Hepatobiliary disorders) | 2 | 2
BILE DUCT OBSTRUCTION (Hepatobiliary disorders) | 2 | 0
BILE DUCT STENOSIS (Hepatobiliary disorders) | 0 | 1
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 1 | 0
HEPATIC FAILURE (Hepatobiliary disorders) | 1 | 0
SEPSIS (Infections and infestations) | 1 | 3
BILIARY TRACT INFECTION (Infections and infestations) | 1 | 0
ESCHERICHIA BACTERAEMIA (Infections and infestations) | 1 | 0
ESCHERICHIA SEPSIS (Infections and infestations) | 1 | 0
LISTERIOSIS (Infections and infestations) | 1 | 0
OSTEOMYELITIS (Infections and infestations) | 1 | 0
PERITONITIS BACTERIAL (Infections and infestations) | 1 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 | 1
HYPERTENSION (Vascular disorders) | 2 | 0
EMBOLISM (Vascular disorders) | 1 | 0
HYPOTENSION (Vascular disorders) | 1 | 0
NECROSIS ISCHAEMIC (Vascular disorders) | 1 | 0
DISEASE PROGRESSION (General disorders) | 0 | 2
NON-CARDIAC CHEST PAIN (General disorders) | 1 | 0
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 1 | 1
MALNUTRITION (Metabolism and nutrition disorders) | 1 | 0
ANAEMIA (Blood and lymphatic system disorders) | 1 | 0
DISSEMINATED INTRAVASCULAR COAGULATION (Blood and lymphatic system disorders) | 1 | 0
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 | 0
EMBOLIC STROKE (Nervous system disorders) | 0 | 1
DELIRIUM (Psychiatric disorders) | 0 | 1
MENTAL STATUS CHANGES (Psychiatric disorders) | 1 | 0
RENAL FAILURE ACUTE (Renal and urinary disorders) | 2 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 1 | 0
SYNOVITIS (Musculoskeletal and connective tissue disorders) | 1 | 0
TUMOUR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cy/GVAX + CRS-207 (N=64) | Cy/GVAX (N=29)
VACCINATION SITE ERYTHEMA (General disorders) | 51 | 25
VACCINATION SITE PRURITUS (General disorders) | 50 | 22
VACCINATION SITE INDURATION (General disorders) | 44 | 23
VACCINATION SITE PAIN (General disorders) | 43 | 20
FATIGUE (General disorders) | 36 | 21
CHILLS (General disorders) | 45 | 8
PYREXIA (General disorders) | 41 | 12
VACCINATION SITE OEDEMA (General disorders) | 22 | 10
VACCINATION SITE HAEMATOMA (General disorders) | 16 | 9
VACCINATION SITE REACTION (General disorders) | 10 | 7
VACCINATION SITE VESICLES (General disorders) | 11 | 6
PAIN (General disorders) | 9 | 4
VACCINATION SITE SWELLING (General disorders) | 7 | 5
ASTHENIA (General disorders) | 7 | 3
VACCINATION SITE NODULE (General disorders) | 8 | 2
INFLUENZA LIKE ILLNESS (General disorders) | 6 | 4
OEDEMA PERIPHERAL (General disorders) | 6 | 2
VACCINATION SITE WARMTH (General disorders) | 5 | 4
VACCINATION SITE HAEMORRHAGE (General disorders) | 3 | 3
CHEST PAIN (General disorders) | 4 | 0
EARLY SATIETY (General disorders) | 3 | 1
NON-CARDIAC CHEST PAIN (General disorders) | 4 | 0
OEDEMA (General disorders) | 2 | 2
VACCINATION SITE DISCOLOURATION (General disorders) | 2 | 1
VACCINATION SITE RASH (General disorders) | 1 | 2
APPLICATION SITE VESICLES (General disorders) | 2 | 0
DISEASE PROGRESSION (General disorders) | 0 | 2
VACCINATION SITE EXFOLIATION (General disorders) | 2 | 0
APPLICATION SITE HAEMATOMA (General disorders) | 1 | 0
APPLICATION SITE PAIN (General disorders) | 1 | 0
CHEST DISCOMFORT (General disorders) | 0 | 1
GAIT DISTURBANCE (General disorders) | 0 | 1
HERNIA (General disorders) | 0 | 1
INFUSION RELATED REACTION (General disorders) | 1 | 0
INJECTION SITE HAEMATOMA (General disorders) | 1 | 0
INJECTION SITE NODULE (General disorders) | 1 | 0
INJECTION SITE PRURITUS (General disorders) | 1 | 0
LOCALISED OEDEMA (General disorders) | 1 | 0
MALAISE (General disorders) | 1 | 0
VACCINATION SITE ESCHAR (General disorders) | 0 | 1
VACCINATION SITE INFLAMMATION (General disorders) | 1 | 0
VACCINATION SITE ULCER (General disorders) | 0 | 1
VENIPUNCTURE SITE THROMBOSIS (General disorders) | 1 | 0
NAUSEA (Gastrointestinal disorders) | 36 | 11
VOMITING (Gastrointestinal disorders) | 30 | 8
ABDOMINAL PAIN (Gastrointestinal disorders) | 19 | 12
CONSTIPATION (Gastrointestinal disorders) | 17 | 8
DIARRHOEA (Gastrointestinal disorders) | 15 | 7
ASCITES (Gastrointestinal disorders) | 10 | 4
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 8 | 3
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 4 | 5
DYSPEPSIA (Gastrointestinal disorders) | 5 | 4
FLATULENCE (Gastrointestinal disorders) | 5 | 1
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 2 | 3
DRY MOUTH (Gastrointestinal disorders) | 4 | 0
GASTRITIS (Gastrointestinal disorders) | 4 | 0
OBSTRUCTION GASTRIC (Gastrointestinal disorders) | 4 | 0
FAECAL INCONTINENCE (Gastrointestinal disorders) | 3 | 0
MELAENA (Gastrointestinal disorders) | 3 | 0
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 1 | 1
DUODENAL ULCER (Gastrointestinal disorders) | 1 | 1
DYSPHAGIA (Gastrointestinal disorders) | 2 | 0
GASTROINTESTINAL SOUNDS (Gastrointestinal disorders) | 1 | 1
ABNORMAL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 2 | 0
LIP BLISTER (Gastrointestinal disorders) | 2 | 0
STOMATITIS (Gastrointestinal disorders) | 2 | 0
ANAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
ANAL PRURITUS (Gastrointestinal disorders) | 1 | 0
COELIAC DISEASE (Gastrointestinal disorders) | 1 | 0
DUODENAL OBSTRUCTION (Gastrointestinal disorders) | 1 | 0
DUODENAL STENOSIS (Gastrointestinal disorders) | 1 | 0
EPIGASTRIC DISCOMFORT (Gastrointestinal disorders) | 1 | 0
EROSIVE OESOPHAGITIS (Gastrointestinal disorders) | 1 | 0
ERUCTATION (Gastrointestinal disorders) | 1 | 0
HAEMORRHOIDS (Gastrointestinal disorders) | 1 | 0
IMPAIRED GASTRIC EMPTYING (Gastrointestinal disorders) | 1 | 0
INTESTINAL PERFORATION (Gastrointestinal disorders) | 1 | 0
MOUTH ULCERATION (Gastrointestinal disorders) | 0 | 1
OESOPHAGEAL DISORDER (Gastrointestinal disorders) | 1 | 0
RETCHING (Gastrointestinal disorders) | 1 | 0
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 | 0
TONGUE DISORDER (Gastrointestinal disorders) | 1 | 0
TOOTHACHE (Gastrointestinal disorders) | 1 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 26 | 10
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 11 | 2
DEHYDRATION (Metabolism and nutrition disorders) | 9 | 2
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 8 | 2
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 8 | 0
HYPOKALAEMIA (Metabolism and nutrition disorders) | 7 | 1
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 8 | 0
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 5 | 2
HYPONATRAEMIA (Metabolism and nutrition disorders) | 7 | 0
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 3 | 1
HYPERKALAEMIA (Metabolism and nutrition disorders) | 2 | 0
CACHEXIA (Metabolism and nutrition disorders) | 1 | 0
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 | 0
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 1 | 0
HYPERMAGNESAEMIA (Metabolism and nutrition disorders) | 1 | 0
IMPAIRED FASTING GLUCOSE (Metabolism and nutrition disorders) | 1 | 0
LACTASE DEFICIENCY (Metabolism and nutrition disorders) | 1 | 0
MALNUTRITION (Metabolism and nutrition disorders) | 1 | 0
METABOLIC ACIDOSIS (Musculoskeletal and connective tissue disorders) | 0 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 13 | 5
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 7 | 3
MYALGIA (Musculoskeletal and connective tissue disorders) | 6 | 4
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 3 | 3
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 3 | 2
NECK PAIN (Musculoskeletal and connective tissue disorders) | 4 | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 5 | 1
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 3 | 1
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 4 | 0
GROIN PAIN (Musculoskeletal and connective tissue disorders) | 1 | 1
NECK MASS (Musculoskeletal and connective tissue disorders) | 2 | 0
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 1
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0
AXILLARY MASS (Musculoskeletal and connective tissue disorders) | 1 | 0
BONE PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 0 | 1
SPINAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0
SYNOVITIS (Musculoskeletal and connective tissue disorders) | 1 | 0
VERTEBRAL COLUMN MASS (Musculoskeletal and connective tissue disorders) | 1 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 18 | 3
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 11 | 2
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 7 | 2
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 3 | 2
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 3 | 2
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 4 | 1
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 2 | 2
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 3 | 1
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 3 | 0
PLEURITIC PAIN (Respiratory, thoracic and mediastinal disorders) | 2 | 1
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 2 | 0
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1 | 1
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 2 | 0
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 2
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 2 | 0
UPPER RESPIRATORY TRACT CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 | 1
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
LARYNGOSPASM (Respiratory, thoracic and mediastinal disorders) | 1 | 0
LUNG INFILTRATION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 1 | 0
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 13 | 2
WEIGHT DECREASED (Investigations) | 9 | 4
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 11 | 0
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 9 | 2
LYMPHOCYTE COUNT DECREASED (Investigations) | 6 | 1
BLOOD BILIRUBIN INCREASED (Investigations) | 5 | 1
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 3 | 2
BLOOD CREATININE INCREASED (Investigations) | 2 | 0
HAEMOGLOBIN DECREASED (Investigations) | 1 | 1
NEUTROPHIL COUNT DECREASED (Investigations) | 2 | 0
WHITE BLOOD CELL COUNT INCREASED (Investigations) | 2 | 0
ACTIVATED PARTIAL THROMBOPLASTIN TIME PROLONGED (Investigations) | 1 | 0
BLOOD ALBUMIN DECREASED (Investigations) | 0 | 1
BLOOD CREATININE (Investigations) | 1 | 0
BLOOD SODIUM DECREASED (Investigations) | 1 | 0
INTERNATIONAL NORMALISED RATIO INCREASED (Investigations) | 1 | 0
LISTERIA TEST POSITIVE (Investigations) | 1 | 0
OXYGEN SATURATION DECREASED (Investigations) | 1 | 0
PLATELET COUNT (Investigations) | 1 | 0
PLATELET COUNT DECREASED (Investigations) | 1 | 0
SKIN TURGOR DECREASED (Investigations) | 0 | 1
TROPONIN I INCREASED (Investigations) | 1 | 0
URINE OUTPUT DECREASED (Investigations) | 1 | 0
URINE OUTPUT INCREASED (Investigations) | 1 | 0
WEIGHT INCREASED (Investigations) | 1 | 0
WHITE BLOOD CELL COUNT (Investigations) | 1 | 0
DIZZINESS (Nervous system disorders) | 14 | 5
HEADACHE (Nervous system disorders) | 6 | 5
SOMNOLENCE (Nervous system disorders) | 9 | 1
DYSGEUSIA (Nervous system disorders) | 3 | 1
BALANCE DISORDER (Nervous system disorders) | 3 | 0
MEMORY IMPAIRMENT (Nervous system disorders) | 3 | 0
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 2 | 1
HYPOAESTHESIA (Nervous system disorders) | 2 | 0
PARAESTHESIA (Nervous system disorders) | 2 | 0
SYNCOPE (Nervous system disorders) | 1 | 1
AMNESIA (Nervous system disorders) | 1 | 0
ANOSMIA (Nervous system disorders) | 1 | 0
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 | 0
COGNITIVE DISORDER (Nervous system disorders) | 0 | 1
EMBOLIC STROKE (Nervous system disorders) | 0 | 1
ENCEPHALOPATHY (Nervous system disorders) | 1 | 0
MENTAL IMPAIRMENT (Nervous system disorders) | 1 | 0
NEURALGIA (Nervous system disorders) | 1 | 0
NEUROPATHY PERIPHERAL (Nervous system disorders) | 1 | 0
SCIATICA (Nervous system disorders) | 1 | 0
SINUS HEADACHE (Nervous system disorders) | 1 | 0
ANAEMIA (Blood and lymphatic system disorders) | 18 | 8
LYMPHOPENIA (Blood and lymphatic system disorders) | 7 | 1
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 4 | 0
NEUTROPENIA (Blood and lymphatic system disorders) | 2 | 1
DISSEMINATED INTRAVASCULAR COAGULATION (Blood and lymphatic system disorders) | 1 | 0
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 1 | 0
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 0 | 1
LYMPH NODE PAIN (Blood and lymphatic system disorders) | 1 | 0
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 1 | 0
HYPOTENSION (Vascular disorders) | 13 | 1
HYPERTENSION (Vascular disorders) | 5 | 3
DEEP VEIN THROMBOSIS (Vascular disorders) | 3 | 2
EMBOLISM (Vascular disorders) | 2 | 1
FLUSHING (Vascular disorders) | 3 | 0
HOT FLUSH (Vascular disorders) | 2 | 0
HAEMATOMA (Vascular disorders) | 1 | 0
NECROSIS ISCHAEMIC (Vascular disorders) | 1 | 0
VENOUS STENOSIS (Vascular disorders) | 1 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 4 | 3
RASH (Skin and subcutaneous tissue disorders) | 6 | 1
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 5 | 0
ALOPECIA (Skin and subcutaneous tissue disorders) | 2 | 1
SKIN HYPERPIGMENTATION (Skin and subcutaneous tissue disorders) | 3 | 0
URTICARIA (Skin and subcutaneous tissue disorders) | 3 | 1
ERYTHEMA (Skin and subcutaneous tissue disorders) | 2 | 0
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 2 | 0
SUBCUTANEOUS NODULE (Skin and subcutaneous tissue disorders) | 1 | 1
COLD SWEAT (Skin and subcutaneous tissue disorders) | 1 | 0
DERMATITIS (Skin and subcutaneous tissue disorders) | 1 | 0
DRY SKIN (Skin and subcutaneous tissue disorders) | 1 | 0
ECCHYMOSIS (Skin and subcutaneous tissue disorders) | 1 | 0
ECZEMA (Skin and subcutaneous tissue disorders) | 1 | 0
HAEMORRHAGE SUBCUTANEOUS (Skin and subcutaneous tissue disorders) | 1 | 0
HYPERKERATOSIS (Skin and subcutaneous tissue disorders) | 1 | 0
ONYCHOMADESIS (Skin and subcutaneous tissue disorders) | 0 | 1
PAIN OF SKIN (Skin and subcutaneous tissue disorders) | 1 | 0
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 0 | 1
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 1 | 0
RASH PRURITIC (Skin and subcutaneous tissue disorders) | 1 | 0
SKIN EXFOLIATION (Skin and subcutaneous tissue disorders) | 1 | 0
INSOMNIA (Psychiatric disorders) | 10 | 2
CONFUSIONAL STATE (Psychiatric disorders) | 3 | 1
DEPRESSION (Psychiatric disorders) | 3 | 1
ANXIETY (Psychiatric disorders) | 2 | 1
DELIRIUM (Psychiatric disorders) | 1 | 2
HALLUCINATION (Psychiatric disorders) | 2 | 0
NIGHTMARE (Psychiatric disorders) | 2 | 0
RESTLESSNESS (Psychiatric disorders) | 2 | 0
AGITATION (Psychiatric disorders) | 0 | 1
DISORIENTATION (Psychiatric disorders) | 1 | 0
MENTAL STATUS CHANGES (Psychiatric disorders) | 1 | 0
TEARFULNESS (Psychiatric disorders) | 1 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 6 | 1
URINARY TRACT INFECTION (Infections and infestations) | 5 | 1
SEPSIS (Infections and infestations) | 2 | 3
NASOPHARYNGITIS (Infections and infestations) | 2 | 0
ORAL HERPES (Infections and infestations) | 2 | 0
BACTERIAL INFECTION (Infections and infestations) | 1 | 0
BILIARY TRACT INFECTION (Infections and infestations) | 1 | 0
BODY TINEA (Infections and infestations) | 0 | 1
CANDIDIASIS (Infections and infestations) | 1 | 0
CLOSTRIDIAL INFECTION (Infections and infestations) | 1 | 0
ESCHERICHIA BACTERAEMIA (Infections and infestations) | 1 | 0
ESCHERICHIA SEPSIS (Infections and infestations) | 1 | 0
HERPES VIRUS INFECTION (Infections and infestations) | 1 | 0
LISTERIOSIS (Infections and infestations) | 1 | 0
LUNG INFECTION (Infections and infestations) | 1 | 0
OESOPHAGEAL CANDIDIASIS (Infections and infestations) | 1 | 0
ORAL INFECTION (Infections and infestations) | 1 | 0
OSTEOMYELITIS (Infections and infestations) | 1 | 0
PENILE INFECTION (Infections and infestations) | 1 | 0
PERITONITIS BACTERIAL (Infections and infestations) | 1 | 0
PNEUMONIA (Infections and infestations) | 0 | 1
SINUSITIS (Infections and infestations) | 1 | 0
URINARY INCONTINENCE (Renal and urinary disorders) | 5 | 0
RENAL FAILURE ACUTE (Renal and urinary disorders) | 3 | 1
CHROMATURIA (Renal and urinary disorders) | 1 | 2
HAEMATURIA (Renal and urinary disorders) | 2 | 0
DYSURIA (Renal and urinary disorders) | 1 | 0
HYDRONEPHROSIS (Renal and urinary disorders) | 1 | 0
INCONTINENCE (Renal and urinary disorders) | 0 | 1
RENAL FAILURE (Renal and urinary disorders) | 0 | 1
URINARY RETENTION (Renal and urinary disorders) | 1 | 0
URINE ODOUR ABNORMAL (Renal and urinary disorders) | 1 | 0
FALL (Injury, poisoning and procedural complications) | 4 | 2
CONTUSION (Injury, poisoning and procedural complications) | 1 | 2
EXCORIATION (Injury, poisoning and procedural complications) | 2 | 0
AVULSION FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
CONCUSSION (Injury, poisoning and procedural complications) | 1 | 0
ESCHAR (Injury, poisoning and procedural complications) | 1 | 0
FOOT FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
GASTROINTESTINAL STOMA COMPLICATION (Injury, poisoning and procedural complications) | 0 | 1
JOINT SPRAIN (Injury, poisoning and procedural complications) | 1 | 0
PATELLA FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
RENAL INJURY (Injury, poisoning and procedural complications) | 0 | 1
RIB FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
SKIN LACERATION (Injury, poisoning and procedural complications) | 1 | 0
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
TOOTH INJURY (Injury, poisoning and procedural complications) | 1 | 0
TRANSFUSION REACTION (Injury, poisoning and procedural complications) | 1 | 0
TACHYCARDIA (Cardiac disorders) | 7 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 1 | 0
BRADYCARDIA (Cardiac disorders) | 1 | 0
CARDIAC DISORDER (Cardiac disorders) | 1 | 0
PERICARDIAL EFFUSION (Cardiac disorders) | 1 | 0
SINUS BRADYCARDIA (Cardiac disorders) | 1 | 0
SINUS TACHYCARDIA (Cardiac disorders) | 1 | 0
CHOLANGITIS (Hepatobiliary disorders) | 3 | 2
BILE DUCT OBSTRUCTION (Hepatobiliary disorders) | 3 | 1
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 3 | 1
BILE DUCT STENOSIS (Hepatobiliary disorders) | 0 | 3
JAUNDICE (Hepatobiliary disorders) | 2 | 0
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 1 | 0
HEPATIC FAILURE (Hepatobiliary disorders) | 1 | 0
VISION BLURRED (Eye disorders) | 3 | 0
BLEPHARITIS (Eye disorders) | 0 | 1
CHROMATOPSIA (Eye disorders) | 1 | 0
CONJUNCTIVAL DISORDER (Eye disorders) | 1 | 0
DRY EYE (Eye disorders) | 1 | 0
IRITIS (Eye disorders) | 0 | 1
PHOTOPSIA (Eye disorders) | 0 | 1
RETINAL TEAR (Eye disorders) | 1 | 0
VITREOUS FLOATERS (Eye disorders) | 1 | 0
EAR DISCOMFORT (Ear and labyrinth disorders) | 3 | 0
CERUMEN IMPACTION (Ear and labyrinth disorders) | 1 | 0
EAR PAIN (Ear and labyrinth disorders) | 1 | 0
TINNITUS (Ear and labyrinth disorders) | 1 | 0
ATROPHIC VULVOVAGINITIS (Reproductive system and breast disorders) | 1 | 0
PELVIC PAIN (Reproductive system and breast disorders) | 1 | 0
PROSTATIC DISORDER (Reproductive system and breast disorders) | 1 | 0
TESTICULAR CYST (Reproductive system and breast disorders) | 1 | 0
VAGINAL DISCHARGE (Reproductive system and breast disorders) | 1 | 0
VULVOVAGINAL PRURITUS (Reproductive system and breast disorders) | 1 | 0
TUMOUR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
HYPERSENSITIVITY (Immune system disorders) | 1 | 0
SEASONAL ALLERGY (Immune system disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less